CLINICAL TRIAL: NCT06077123
Title: Differential Effects of a Telemonitoring Platform in the Development of Chemotherapy-Associated Toxicity: A Randomised Trial
Brief Title: Telemonitoring Platforms and Chemotherapy-Associated Toxicity
Acronym: DETECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Andres Bello (Other)
Collaborators: Centro para la Prevención y Control del Cáncer (CECAN), Santiago, Chile (Unknown)
Responsible Party: Principal Investigator, Felipe Martinez Lomakin, Associate Professor, Universidad Nacional Andres Bello
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UNAB-004
Record Dates: First submitted 2023-10-04; First posted 2023-10-11 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Cancer; Chemotherapeutic Agent Toxicity
Keywords: Telemonitoring; Internet; Smartphones; Quality of Life; User Satisfaction
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio using a permuted block method to receive one of the two intervention strategies.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemonitoring Platform (Experimental): Patients allocated to the active intervention group will receive a smartphone application called Contigo. This tool aims to detect signs and symptoms of oncology drug toxicity and delivering educational content that enables the patient to have tools to address common clinical situations associated with the diagnosis and treatment of their disease.
  Interventions: Device: Contigo Application
- Traditional Follow-Up (No Intervention): Those assigned to the traditional follow-up group will receive standard care and in-person check-ups as determined by their attending physician.

INTERVENTIONS:
Device: Contigo Application — Contigo, a smartphone application, aims to achieve two main objectives: monitoring cancer patients for early detection of oncology drug toxicity signs and providing educational content to empower patients in handling clinical challenges tied to their diagnosis and treatment. Monitoring involves modules and sub-modules where patients input experiences through oncology-related questionnaires. Weekly checks for chemotherapy toxicity-associated symptoms use a validated questionnaire (PRO-CTCAE). Severe toxicity triggers immediate alerts, while milder cases receive educational guidance. Data collected is shared with healthcare providers. Educational health content has been created by professionals, encompassing cancer-specific topics, healthcare processes, administration, health coverage, self-awareness, and self-care practices. The content is based on scientific evidence, official reports, and group sessions involving healthcare professionals and cancer patients.
  Arms: Telemonitoring Platform

SUMMARY:
The primary objective of this trial is to evaluate the impact of a telemonitoring platform on patient satisfaction with care amongst adult cancer patients receiving chemotherapy. The key questions it seeks to address revolve around the potential improvements in both quality of life and satisfaction with healthcare. Participants in the trial will be provided with a specialized application developed by a team of experienced oncology professionals. Their quality of life and healthcare experience will be compared with that of the control group, who will only receive the standard in-person check-ups established by their healthcare team.

DETAILED DESCRIPTION:
This protocol describes a randomized parallel-group clinical trial among recently diagnosed patients with solid carcinomas preparing for curative intent chemotherapy at Hospital Sótero del Río and UC-Christus Health Network centers. Eligible adult patients (>18 years) diagnosed with lung, gastric, gallbladder, colon, breast, or cervical carcinoma, scheduled for outpatient curative intent chemotherapy within UC-Christus Health Network or Hospital Sotero del Rio from November 2023 to July 2024, proficient in Spanish, and possessing a smartphone (iOS® or Android®) will be recruited. Exclusions include those undergoing concomitant radiotherapy, sensory impairments hindering app use, cognitive or psychiatric issues, and unwillingness to participate. Participants will be randomized 1:1 to receive either the Contigo smartphone application or standard care. Contigo aims to monitor chemotherapy toxicity symptoms and deliver cancer-related educational content. The application includes modules addressing cancer care, self-perception of health, patient experiences, frequently asked questions, community resources, and scheduling. Information collected by the app will be available to healthcare providers. Patients will receive the app for free and undergo training on its usage. Weekly toxicity assessments using Patient-Reported Outcomes of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) will be conducted. The control group will receive standard in-person care. The primary outcome is patient experience during chemotherapy, measured using the OUT-PATSAT-35 questionnaire three months after randomization. Secondary outcomes include severe chemotherapy-associated toxicity, quality of life, and user satisfaction with the application. A sample size of 80 participants (40 per group) was calculated. Descriptive analysis will utilize means, standard deviation, frequencies, and percentages. Inferential analysis will involve t-tests, Mann-Whitney U tests, Fisher's Exact Test, and Kaplan-Meier survival curves. All analyses will adhere to intention-to-treat principles and use Stata v.16.0® software. No subgroup analyses have been programmed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years)
* Histologically confirmed diagnosis of lung, gastric, gallbladder, colon, breast, or cervical carcinoma in any of its forms and stages
* Initiating an outpatient curative intent chemotherapy regimen within the facilities of UC-Christus Health Network or Hospital Sotero del Río during the months of November 2023 to July 2024
* Proficient in the Spanish language
* Possess a smartphone, regardless of the native operating system (iOS® or Android®)

Exclusion Criteria:

* Individuals undergoing concomitant radiotherapy
* Those with any form of sensory impairment hindering the use of the application
* Those with cognitive impairment or psychiatric pathology preventing the use of the application
* Those who do not wish to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Patient Experience Scores | 3 months after randomization
  Patient Satisfaction with Healthcare Services Provided using the European Organisation for Research and Treatment of Cancer Satisfaction with Cancer Care for Outpatients questionnaire (EORTC OUTPATSAT-35). Scores can range from 0 to 100 points, with higher scores implying greater satisfaction with care.

SECONDARY OUTCOMES:
Quality of Life Scores | 3 months after randomization
  Quality of Life scores as assessed by the EuroQol 5 Dimension (EQ-5D) questionnaire. The index score ranges from 0 to 1, with higher values indicating an overall better quality of life.
Severe adverse event attributable to chemotherapy | 3 months after randomization
  Proportion of patients who develop a severe adverse event attributable to cytotoxic chemotherapy. Severe events will be those of grade 3 to 5 of the Common Terminology Criteria for Adverse Events classification.
Hospitalizations due to a chemotherapy adverse event | 3 months after randomization
  Propotion of patients who require hospitalizations due to an adverse event attributable to cytotoxic chemotherapy
Chemotherapy dose adjustment | 3 months after randomization
  Proportion of patients who require a reduction in their chemotherapy dose in each group.
Emergency department visits | 3 months after randomization
  Median number of emergency department visits in each study group

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Nervi, MD, Study Chair — Pontificia Universidad Catolica de Chile; Manuel Espinoza, PhD, Principal Investigator — Pontificia Universidad Catolica de Chile; Carla Taramasco, PhD, Study Director — Escuela de Ingeniería, Universidad Andrés Bello
Locations (2):
- Chile (2):
  - Centro del Cáncer, Pontificia Universidad Católica de Chile, Santiago
  - Complejo Asistencial Dr. Sotero del Río, Santiago

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized individual participant data including clinical characteristics and outcomes will be made available to other researchers on reasonable request, such as to inform the conduction a systematic review on telemonitoring platforms for providing care to patients with cancers.

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Arnold B, Mitchell SA, Lent L, Mendoza TR, Rogak LJ, Barragan NM, Willis G, Medina M, Lechner S, Penedo FJ, Harness JK, Basch EM; PRO-CTCAE Spanish Translation and Linguistic Validation Study Group. Linguistic validation of the Spanish version of the National Cancer Institute's Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). Support Care Cancer. 2016 Jul;24(7):2843-51. doi: 10.1007/s00520-015-3062-5. Epub 2016 Feb 2. PMID 26838022
- [Background] Basch E, Stover AM, Schrag D, Chung A, Jansen J, Henson S, Carr P, Ginos B, Deal A, Spears PA, Jonsson M, Bennett AV, Mody G, Thanarajasingam G, Rogak LJ, Reeve BB, Snyder C, Kottschade LA, Charlot M, Weiss A, Bruner D, Dueck AC. Clinical Utility and User Perceptions of a Digital System for Electronic Patient-Reported Symptom Monitoring During Routine Cancer Care: Findings From the PRO-TECT Trial. JCO Clin Cancer Inform. 2020 Oct;4:947-957. doi: 10.1200/CCI.20.00081. PMID 33112661
- [Background] Zarate V, Kind P, Valenzuela P, Vignau A, Olivares-Tirado P, Munoz A. Social valuation of EQ-5D health states: the Chilean case. Value Health. 2011 Dec;14(8):1135-41. doi: 10.1016/j.jval.2011.09.002. Epub 2011 Nov 6. PMID 22152184
- [Background] Arraras JI, Illarramendi JJ, Viudez A, Lecumberri MJ, de la Cruz S, Hernandez B, Zarandona U, Bredart A, Martinez M, Salgado E, Lainez N, Vera R. The cancer outpatient satisfaction with care questionnaire for chemotherapy, OUT-PATSAT35 CT: a validation study for Spanish patients. Support Care Cancer. 2012 Dec;20(12):3269-78. doi: 10.1007/s00520-012-1467-y. Epub 2012 May 2. PMID 22549507
- [Derived] Martinez F, Taramasco C, Espinoza M, Acevedo J, Goic C, Nervi B. Differential Effects of a Telemonitoring Platform in the Development of Chemotherapy-Associated Toxicity: A Randomized Trial Protocol. Diagnostics (Basel). 2024 Mar 14;14(6):619. doi: 10.3390/diagnostics14060619. PMID 38535039
- See also: Center for Cancer Control and Prevention Website — https://cecan.cl/